CLINICAL TRIAL: NCT05349071
Title: Preoperative Methylprednisolone on Thoracic Endovascular Repair for Reducing Post-implantation Syndrome
Brief Title: PreOperative Methylprednisolone on Thoracic Endovascular Repair for Reducing Post-implantation Syndrome (POMTEVAR)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Guangdong Provincial People's Hospital (Other)
Collaborators: The First Affiliated Hospital of Guangzhou Medical University (Other); Shenzhen People's Hospital (Other)
Responsible Party: Principal Investigator, Jianfang Luo, chief physician, Guangdong Provincial People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: KY-Z-2021-581-02
Record Dates: First submitted 2022-04-21; First posted 2022-04-27 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Methylprednisolone; Thoracic Endovascular Repair; Post-implantation Syndrome; Type B Aortic Dissection
Keywords: type B aortic dissection; post-implantation syndrome; thoracic endovascular repair; methylprednisolone
MeSH Terms: interventions — Methylprednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- methylprednisolone group (Experimental): a single preoperative dose of 500 mg of methylprednisolone diluted in 250 mL of physiological saline 2 hours before surgery as a 30-minute infusion.
  Interventions: Drug: methylprednisolone
- physiological saline group (Active Comparator): a single preoperative dose of 250 mL of physiological saline 2 hours before surgery as a 30-minute infusion.
  Interventions: Drug: physiological saline

INTERVENTIONS:
Drug: methylprednisolone — a single preoperative dose of 500 mg of methylprednisolone diluted in 250 mL of physiological saline 2 hours before surgery as a 30-minute infusion.
  Arms: methylprednisolone group
Drug: physiological saline — a single preoperative dose of 250 mL of physiological saline 2 hours before surgery as a 30-minute infusion.
  Arms: physiological saline group

SUMMARY:
POMTEVAR trial is a multicenter, open-label and prospective random controlled study. Approximately 158 patients will be randomly allocated to thoracic endovascular repair (TEVAR) alone group or TEVAR plus methylprednisolone group and managed with respective treatment strategies. All study patients will be followed up in the outpatient clinic and undergo CT scans after 3 months from randomization. The primary objective is to test the hypothesis that PIS is lower in TEVAR plus methylprednisolone group than that in TEVAR alone group. The secondary objective is to test the hypothesis that changes of postoperative inflammatory indicators, incidence of postoperative acute renal failure and postoperative delirium, postoperative pain score are lower in TEVAR plus methylprednisolone group than that in TEVAR alone. In addition, 3-month all-cause death, 3-month major adverse cardiovascular events, 3-month aorta-related adverse events and 3-month aortic remodeling are compared between groups.

DETAILED DESCRIPTION:
POMTEVAR trial is a multicenter, open-label and prospective random controlled study. Approximately 158 patients will be randomly allocated to thoracic endovascular repair (TEVAR) alone group or TEVAR plus methylprednisolone group and managed with respective treatment strategies. All study patients will be followed up in the outpatient clinic and undergo CT scans after 3 months from randomization.

The primary objective is to test the hypothesis that PIS is lower in TEVAR plus methylprednisolone group than that in TEVAR alone group. The secondary objective is to test the hypothesis that changes of postoperative inflammatory indicators, incidence of postoperative acute renal failure and postoperative delirium, postoperative pain score are lower in TEVAR plus methylprednisolone group than that in TEVAR alone. In addition, 3-month all-cause death, 3-month major adverse cardiovascular events, 3-month aorta-related adverse events and 3-month aortic remodeling are compared between groups.

TEVAR plus glucocorticoids group: Patients receive a single preoperative dose of 500 mg of methylprednisolone diluted in 250 mL of physiological saline 2 hours before TEVAR as a 30-minute infusion.

TEVAR alone group: Patients receive a single preoperative dose of 250 mL of physiological saline 2 hours before TEVAR as a 30-minute infusion.

TEVAR steps:According to the preoperative imaging, the potential risk location of the aortic dissection or rupture and the extent of lesion involvement are evaluated, and the appropriate anchoring zone is selected to ensure a sufficient anchorage area of more than 15 mm. If the distance between the potential accident site and the left subclavian artery (LSA) is less than 15 mm, LSA will be covered to obtain sufficient anchoring area. LSA revascularization will be performed by chimney technique or hybrid operation, depending on the choice of the surgeon. The left femoral artery is punctured or cut, the 5F artery sheath is inserted, and the pigtail catheter is inserted into the ascending aorta along the sheath. Next, the aortic covered stent was implanted reverse through the femoral artery under the guidance of the wire. When the stent was released, rapid pacing or intravenous antihypertensive drugs was used to ensure that the blood pressure was lower than 90 mmHg. After stent implantation, re-angiography to confirm the stent location and blood flow, which will indicate whether the operation was successful or not. After all above, the patients will be observed in hospital for at least 3 days. Controls of the blood pressure and heart rate and relief of the symptoms will meet the discharge criteria.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years;
2. Be confirmed as Stanford type B aortic dissection by aorta computed tomography;
3. From onset to first clinical attach <90 days;
4. The subject or legal guardian understands the nature of the study and agrees to its provisions on a written informed consent form;
5. Availability for the appropriate follow-up visits during the follow-up period;
6. Capability to follow all study requirements.

Exclusion Criteria:

1. Laboratory examination in the last 3 months suggested severe renal dysfunction (serum creatinine >176.8umol/L or estimated creatinine clearance eGFR <30ml/min;
2. Laboratory examination in the last 3 months suggested severe liver dysfunction (ALT> 2x Max or TBIL> 2x Max);
3. Diabetics with poor glycemic control: fasting blood glucose ≥13.9mmol/L or hBA1c ≥8.5%;
4. Severe hypokalemia (Serum potassium ion concentration was less than 2.5mmol/L);
5. HIV positive, hepatitis B or C positive;
6. Immune inflammatory diseases (except skin and respiratory diseases that can be treated locally);
7. Glaucoma;
8. Gastric or duodenal ulcer;
9. Active infection (persisting body temperature >38℃; etiological evidence or imaging evidence);
10. On immunosuppressive therapy;
11. Patients with malignant tumor whose life expectancy is less than 1 year;
12. Genetic diseases, including Turner syndrome, Marfan syndrome, Ehlers-Danlos syndrome, Loeys-Dietz syndrome and other connective tissue diseases;
13. Rheumatic immune diseases, including multiple arteritis, giant cell arteritis, polyarteritis nodosum, etc;
14. Pregnant women;
15. Severe mental illness;
16. Poor compliance, difficult to cooperate with follow-up;
17. Participate in another investigationdrug or medical device study or another investigationstudy of an approved drug or medical device within 30 days prior to the first visit of the current study;
18. Any conditions or laboratory findings that the investigator considers inappropriate for inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Estimated)
Dates: Start 2022-05-01 (Estimated); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Rate of post-implantation syndrome | the first 5 postoperative days
  the incidence of post-implantation syndrome in the first 5 postoperative days

SECONDARY OUTCOMES:
Rate of acute renal failure | the first 5 postoperative days
  the rate of acute renal failure in the first 5 postoperative days
Rate of postoperative delirium | the first 5 postoperative days
  the rate of postoperative delirium in the first 5 postoperative days
postoperative pain score | 1 hour and 24 hours after thoracic endovascular repair
  postoperative pain score
Rate of all-cause mortality | three months
  All-cause mortality includes aortic-related and nonaortic-related mortality
Rate of aortic-related mortality | three months
  Aortic-related death was defined as death attributable to an aortic cause during the initial admission or follow-up
Incidence of re-intervention | three months
  secondary intervention
Incidence of major adverse cardiovascular events | three months
  cardiac death, non-fatal acute myocardial infarction (ST and non-ST), ischemic stroke or transient ischemic attack
Incidence of aorta-related adverse events | three months
  aortic rupture, aortic-related death, re-intervention and paraplegia

CONTACTS AND LOCATIONS:
Overall Officials: Jianfang Luo, MD, Study Chair — Guangdong Provincial People's Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Erbel R, Aboyans V, Boileau C, Bossone E, Bartolomeo RD, Eggebrecht H, Evangelista A, Falk V, Frank H, Gaemperli O, Grabenwoger M, Haverich A, Iung B, Manolis AJ, Meijboom F, Nienaber CA, Roffi M, Rousseau H, Sechtem U, Sirnes PA, Allmen RS, Vrints CJ; ESC Committee for Practice Guidelines. 2014 ESC Guidelines on the diagnosis and treatment of aortic diseases: Document covering acute and chronic aortic diseases of the thoracic and abdominal aorta of the adult. The Task Force for the Diagnosis and Treatment of Aortic Diseases of the European Society of Cardiology (ESC). Eur Heart J. 2014 Nov 1;35(41):2873-926. doi: 10.1093/eurheartj/ehu281. Epub 2014 Aug 29. No abstract available. PMID 25173340
- [Background] Bossone E, LaBounty TM, Eagle KA. Acute aortic syndromes: diagnosis and management, an update. Eur Heart J. 2018 Mar 1;39(9):739-749d. doi: 10.1093/eurheartj/ehx319. PMID 29106452
- [Background] Evangelista A, Isselbacher EM, Bossone E, Gleason TG, Eusanio MD, Sechtem U, Ehrlich MP, Trimarchi S, Braverman AC, Myrmel T, Harris KM, Hutchinson S, O'Gara P, Suzuki T, Nienaber CA, Eagle KA; IRAD Investigators. Insights From the International Registry of Acute Aortic Dissection: A 20-Year Experience of Collaborative Clinical Research. Circulation. 2018 Apr 24;137(17):1846-1860. doi: 10.1161/CIRCULATIONAHA.117.031264. PMID 29685932
- [Background] Liu D, Luo H, Lin S, Zhao L, Qiao C. Comparison of the efficacy and safety of thoracic endovascular aortic repair with open surgical repair and optimal medical therapy for acute type B aortic dissection: A systematic review and meta-analysis. Int J Surg. 2020 Nov;83:53-61. doi: 10.1016/j.ijsu.2020.08.051. Epub 2020 Sep 11. PMID 32927144
- [Background] Li FR, Wu X, Yuan J, Wang J, Mao C, Wu X. Comparison of thoracic endovascular aortic repair, open surgery and best medical treatment for type B aortic dissection: A meta-analysis. Int J Cardiol. 2018 Jan 1;250:240-246. doi: 10.1016/j.ijcard.2017.10.050. Epub 2017 Oct 16. PMID 29066151
- [Background] De La Motte L, Vogt K, Panduro Jensen L, Groenvall J, Kehlet H, Veith Schroeder T, Lonn L. Incidence of systemic inflammatory response syndrome after endovascular aortic repair. J Cardiovasc Surg (Torino). 2011 Feb;52(1):73-9. PMID 21224813
- [Background] Zhu Y, Luo S, Ding H, Liu Y, Huang W, Xie N, Li J, Xue L, Luo J. Predictors associated with an increased prevalence of postimplantation syndrome after thoracic endovascular aortic repair for type B aortic dissectiondagger. Eur J Cardiothorac Surg. 2019 May 1;55(5):998-1005. doi: 10.1093/ejcts/ezy379. PMID 30521031
- [Background] Arnaoutoglou E, Papas N, Milionis H, Kouvelos G, Koulouras V, Matsagkas MI. Post-implantation syndrome after endovascular repair of aortic aneurysms: need for postdischarge surveillance. Interact Cardiovasc Thorac Surg. 2010 Oct;11(4):449-54. doi: 10.1510/icvts.2010.242628. Epub 2010 Jul 19. PMID 20643821
- [Background] Belkin N, Jackson BM, Foley PJ, Damrauer SM, Kalapatapu V, Golden MA, Fairman RM, Kelz RR, Wang GJ. Length of Stay after Thoracic Endovascular Aortic Repair Depends on Indication and Acuity. Ann Vasc Surg. 2019 Feb;55:157-165. doi: 10.1016/j.avsg.2018.06.027. Epub 2018 Sep 11. PMID 30217710
- [Background] Chan TCW, Cheung CW, Wong SSC, Chung AYF, Irwin MG, Chan PK, Fu H, Yan CH, Chiu KY. Preoperative dexamethasone for pain relief after total knee arthroplasty: A randomised controlled trial. Eur J Anaesthesiol. 2020 Dec;37(12):1157-1167. doi: 10.1097/EJA.0000000000001372. PMID 33105245
- [Background] de la Motte L, Kehlet H, Vogt K, Nielsen CH, Groenvall JB, Nielsen HB, Andersen A, Schroeder TV, Lonn L. Preoperative methylprednisolone enhances recovery after endovascular aortic repair: a randomized, double-blind, placebo-controlled clinical trial. Ann Surg. 2014 Sep;260(3):540-8; discussion 548-9. doi: 10.1097/SLA.0000000000000895. PMID 25115430
- [Background] Nienaber CA, Clough RE, Sakalihasan N, Suzuki T, Gibbs R, Mussa F, Jenkins MP, Thompson MM, Evangelista A, Yeh JS, Cheshire N, Rosendahl U, Pepper J. Aortic dissection. Nat Rev Dis Primers. 2016 Jul 21;2:16053. doi: 10.1038/nrdp.2016.53. PMID 27440162
- [Background] Czerny M, Schmidli J, Adler S, van den Berg JC, Bertoglio L, Carrel T, Chiesa R, Clough RE, Eberle B, Etz C, Grabenwoger M, Haulon S, Jakob H, Kari FA, Mestres CA, Pacini D, Resch T, Rylski B, Schoenhoff F, Shrestha M, von Tengg-Kobligk H, Tsagakis K, Wyss TR; EACTS/ESVS scientific document group. Current options and recommendations for the treatment of thoracic aortic pathologies involving the aortic arch: an expert consensus document of the European Association for Cardio-Thoracic surgery (EACTS) and the European Society for Vascular Surgery (ESVS). Eur J Cardiothorac Surg. 2019 Jan 1;55(1):133-162. doi: 10.1093/ejcts/ezy313. No abstract available. PMID 30312382
- [Background] Polderman JA, Farhang-Razi V, Van Dieren S, Kranke P, DeVries JH, Hollmann MW, Preckel B, Hermanides J. Adverse side effects of dexamethasone in surgical patients. Cochrane Database Syst Rev. 2018 Nov 23;11(11):CD011940. doi: 10.1002/14651858.CD011940.pub3. PMID 30480776